CLINICAL TRIAL: NCT06683313
Title: Comparison of the Combination of Popliteal Sciatic and Femoral Block With the Combination of Ipack Adductor Canal Block Duration in Elective Knee Surgeries
Brief Title: Comparison of the Combination of Popliteal Sciatic and Femoral Block With the Combination of Ipack Adductor Canal Blocks
Acronym: kneesurgery
Status: Completed | Type: Observational
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Responsible Party: Principal Investigator, Döndü Genc Moralar, associate professor, Gaziosmanpasa Research and Education Hospital
Other Study IDs: knee surgeries blocks
Record Dates: First submitted 2024-11-08; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Post-operative Analgesia; Early Mobility
Keywords: femoral block; knee surgery; sciatic nerve block; IPACK block; Adductor Canal Block; post-operative analgesia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- adductor canal block add ipack: Patients who received ipack add femoral canal block for postoperative analgesia
  Interventions: Combination Product: combination adductor canal and IPACK block
- femoral block add popliteal sciatic: Patients who underwent popliteal sciatic block add femoral block for postoperative analgesia
  Interventions: Combination Product: combination femoral nerve and popliteal sciatica block

INTERVENTIONS:
Combination Product: combination femoral nerve and popliteal sciatica block — Combination of femoral nerve and popliteal sciatica block performed after knee surgery
  Other Names: group FS
  Groups: femoral block add popliteal sciatic
Combination Product: combination adductor canal and IPACK block — Combination of adductor canal and IPACK block performed after knee surgery
  Other Names: group AI
  Groups: adductor canal block add ipack

SUMMARY:
Comparison of the combination of popliteal sciatic and femoral block with the combination of ipack adductor canal blocks and mobilization and analgesia duration in elective knee surgeries

DETAILED DESCRIPTION:
There is concern that about half of patients with elective knee surgery report severe knee pain immediately after surgery. Optimal postoperative knee analgesia is important not only for patient comfort and satisfaction, but also to accelerate mobilization, functional recovery, and hospital discharge. To facilitate earlier ambulation and provide superior pain control, while striving for shorter hospital stays and same-day discharge for patients There is an increasing emphasis on multimodal analgesia and motor sparing regional anesthesia blocks.

To compare the postoperative analgesic efficacy of ipack adductor canal and femoral popliteal sciatic blocks in elective knee surgeries, and the first mobilization (bromage 0) times of motor block after spinal anesthesia. Our primary aim is to compare the ipack adductor canal block added after spinal anesthesia in elective knee surgeries with the combination of femoral + popliteal sciatic block. post of blocks To evaluate the operative mobilization (bromage 0) and analgesia times. Our secondary aims are to evaluate the first 4, 8, 12, 24 hours VAS (visual analog scale) values, first analgesia time, post op 1 hour bromage scores, postoperative nausea, vomiting, and discharge times, side effects. compare the incidence of effects.

ELIGIBILITY:
Inclusion Criteria: knee operation,

-

Exclusion Criteria:Patients who did not consent to the procedure, those with coagulopathy, a known allergy to local anesthetics, a BMI > 35 kg/m², chronic analgesic and opioid use, mental or psychiatric disorders, or inability -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 to 75 who will undergo knee surgery
Sampling Method: Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
postoperative first mobilization time | 24 hour
  After receiving spinal anesthesia, patients undergoing elective knee surgery were taken to the operating room. Postoperatively, patients were randomly assigned into two groups using a closed-envelope method. In the first group, patients in the supine position received an adductor canal block with 20 ml of 0.025% bupivacaine and an IPACK block with an additional 20 ml of 0.025% bupivacaine. In the second group, patients in the supine position received a femoral nerve block with 20 ml of 0.025% bupivacaine and a sciatic nerve block administered via the popliteal region with an additional 20 ml of 0.025% bupivacaine. Motor block, analgesia, and mobilization times were assessed at the 2nd, 4th, 8th, and 24th hours postoperatively.In the postoperative period, patients' motor functions were assessed at specific intervals (e.g., at the 2nd, 4th, 8th, 12th and 24th hours) using the Bromage Scale. During each assessment, patients were asked to move their hip, knee, and ankle joints.

SECONDARY OUTCOMES:
Numerical Rating Scale (NRS) Scores | 24 hour
  NRS scores were evaluated at the 2nd, 4th, 8th, 12th, and 24th hours. The Numerical Rating Scale (NRS) is a pain assessment tool where patients rate their pain intensity on a scale from 0 to 10, with 0 indicating no pain and 10 representing the worst pain imaginable.

CONTACTS AND LOCATIONS:
Overall Officials: osman çelik, Principal Investigator — Gaziosmanpasa Research and Education Hospital
Locations (1):
- Gaziosmanpasa Research and Education Hospital, Istanbul, 34000, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
It will be shared upon request from the corresponding author via email if desired.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 2 year
Access Criteria: Those who are healthcare professionals